CLINICAL TRIAL: NCT05764746
Title: Can Triple Artemisinin-based Combination Therapy for Treatment of Uncomplicated Plasmodium Falciparum Malaria, Delay Drug Resistance Development of Plasmodium Falciparum in Tanzania: a Randomized Three Arm Clinical Trial
Brief Title: Triple Artemisinin-based Combination Therapy for Delaying Drug Resistance Development - a Randomized Clinical Trial
Acronym: 3ACT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Muhimbili University of Health and Allied Sciences (Other)
Collaborators: The Swedish Research Council (Other Government); Uppsala University (Other)
Responsible Party: Principal Investigator, Billy Ngasala, Associate Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3ACT-2023
Record Dates: First submitted 2023-02-01; First posted 2023-03-13 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-04

CONDITIONS: Uncomplicated Plasmodium Falciparum Malaria
Keywords: Artemisinin-based Combination Therapy; Plasmodium falciparum; Uncomplicated malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: A health facility-based, three-arm partially blinded randomized clinical trial will be conducted to assess efficacy and safety of a sequential administration of artemether-lumefantrine followed immediately by artesunate-amodiaquine (AL+ASAQ) or artemether-lumefantrine with by amodiaquine (AL+AQ) compared to artemether-lumefantrine plus placebo (AL+PBO).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Artemether-lumefantrine followed by artesunate amodiaquine (Experimental): a standard 3-days dosage, twice a day course of Artemether-Lumefantrine (20/120mg) immediately followed by a standard 3-days, once a day course of Artesunate-Amodiaquine (40base)
  Interventions: Drug: Artemether-lumefantrine then Artesunate amodiaquine
- Artemether-lumefantrine with Amodiaquine (Experimental): a standard 3-days dosage of Artemether-Lumefantrine (20/120mg) given together with Amodiaquine hydrocloride(40 base) followed by placebo for another 3 days;
  Interventions: Drug: Artemether-lumefantrine and Amodiaquine Drug Combination
- Artemether-Lumefantrine alone (Active Comparator): a standard 3-days dosage of Artemether-Lumefantrine (20/120mg) followed by placebo for another 3 days
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Artemether-lumefantrine and Amodiaquine Drug Combination — AL and AQ will be given together for three days then followed by placebo for three days
  Other Names: AL+AQ
  Arms: Artemether-lumefantrine with Amodiaquine
Drug: Artemether-lumefantrine then Artesunate amodiaquine — AL will be given twice a day for three days then followed by artesunate amodiaquine once a day for three days
  Other Names: AL then ASAQ
  Arms: Artemether-lumefantrine followed by artesunate amodiaquine
Drug: Artemether-lumefantrine — This will be the comparator arm as standard treatment, where only AL will be given twice a day for three days then placebo for three days
  Other Names: AL + Placebo
  Arms: Artemether-Lumefantrine alone

SUMMARY:
Background: Artemisinin resistance has emerged in parts of Southeast Asia, and there are reports in Africa of reduced susceptibility of Plasmodium falciparum parasites against artemisinin-based combination therapy (ACT). No new drugs are available in the pipeline to replace ACTs in case they fail.

This study aims to assess whether a sequential administration of triple ACTs with different partner-drugs can improve the efficacy of ACT for treatment of uncomplicated malaria.

Methods: A health facility-based, three-arm partially blinded randomized clinical trial will be conducted to assess efficacy and safety of a sequential administration of artemether-lumefantrine followed immediately by artesunate-amodiaquine (AL+ASAQ) or artemether-lumefantrine with by amodiaquine (AL+AQ) compared to artemether-lumefantrine plus placebo (AL+PBO). Eligible children aged 6 - 120 months and with microscopy confirmed uncomplicated P. falciparum malaria will be enrolled, administered with trial medicines and followed-up at 0 (just prior to first drug intake) and 8 hours on day 0, 12 hourly on days 1, 2, 3, 4, 5, followed by once daily on days 6, 7, 8, 9, 10, 11, 12, 13, 14, 21, 28, 35, 42 and 56 for clinical and laboratory evaluations. Clinical evaluation will involve assessment of signs and symptoms related to the disease and or trial medicine during follow-up. Laboratory evaluation will include microscopic determination of presence of malaria parasites and species, hemoglobin level, molecular analysis for markers of drug resistance and to differentiate recrudescence from new infection. The primary outcome will be Polymerase Chain Reaction (PCR)-adjusted adequate clinical and parasitological cure rate on days 28 and 42.

Expected outcomes: The findings will give an insight on whether 3 ACTs are more efficacious than the use of first-line regimen alone, and are tolerable for treatment of uncomplicated falciparum malaria.

ELIGIBILITY:
Patients presenting at the health facility with suspected acute uncomplicated malaria will be screened for eligibility.

Inclusion Criteria:

* Age from 6 - 120 months
* Weight ≥ 5 kg
* Body temperature ≥37.5°C or history of fever in the last 24 hours
* Microscopy confirmed P. falciparum mono-infection
* Parasitemia level of 1000-200000/μL
* Ability to swallow oral medication
* Ability and willingness to abide by the study protocol and the stipulated follow-up visits
* A written proxy informed consent from a parent/guardian

Exclusion Criteria:

* Children aged below 6 months will not be included in the study because ACTs are contraindicated in this group.
* Evidence of severe malaria or danger signs
* Known allergy to trial medicines
* Reported antimalarial intake ≤2 weeks
* Haemoglobin <5 g/dL
* Blood transfusion within last 90 days
* Febrile condition other than malaria
* Known underlying chronic or severe disease (including severe malnutrition).

Ages: 6 Months to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 384 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Crude recurrent parasitemia by day 56 in the respective arms | 56th day since enrolment
  Laboratory assessment of parasitemia using light microscopy performed at last day of follow up will be the primary outcome assessing the differences in proportion of patients with recurrent parasitemia.

SECONDARY OUTCOMES:
PCR adjusted cure rates by day 28, 42 and 56. | Through study completion, an average of 1 year
  Assessment of cure rate as determined by parasitemia to distinguish recrudescence and reinfections

OTHER OUTCOMES:
Median time to recurrent parasitemia by microscopy | 56 days since enrolment
  This outcome compares across the three arms how long it takes until patients return with parasitemia. It will provide information on the post treatment prophylaxis of each arm.
PCR determined parasite clearance times | Baseline to day 3
  PCR determined parasite clearance times are determined by using PCR to measure the amount of parasite DNA in the patient's blood at various time points after treatment. The parasite clearance time is then calculated as the time it takes for the amount of parasite DNA to fall below a certain threshold level, indicating that the parasite has been cleared from the patient's blood.
Maximum plasma concentrations (Cmax) of the intervention drugs. | Baseline and Day 7
  The Pharmacokinetics profiles of artesunate/dihydroartemisinin, lumefantrine/desbutyl-lumefantrine and amodiaquine/desethyl-amodiaquine will be assessed, focusing on Plasma concentrations to determine Cmax.
Change in hemoglobin level (g/dl) | Baseline and day 7
  Haemoglobin concentration will be measured at baseline day 0 on day 7 to determine whether patients are anemic or not. . Anemia will be categorized as mild (Hb < 11 g/dL), moderate (< 7 g/dL) or severe (Hb < 5 g/dL).
Proportion of Microscopy determined gametocyte carriage | Baseline and day 3
  Assessment of how many patients in each treatment arm harbour gametocytes
Prevalence of genetic markers of drug resistance. | Through study completion, an average of 1 year
  Selection of genetic markers of drug resistance among recurrent parasitemia during follow-up and during the early treatment phase. The markers will include P. falciparum chloroquine resistance transporter gene (Pfcrt), and P. falciparum multidrug resistance gene 1 (Pfmdr1) for lumefantrine and amodiaquine; P. falciparum multidrug resistance proteins, the sarco/endoplasmic reticulum Ca2+-ATPase orthologue of P. falciparum (pfatp6), and P. falciparum kelch propeller gene 13 (PfKelch13) for artemisinin; and plasmepsin 2 and 3 for piperaquine.

CONTACTS AND LOCATIONS:
Overall Officials: Billy E Ngasala, PhD, Principal Investigator — Muhimbili University of Health and Allied Sciences; Andreas Mårtensson, PhD, Principal Investigator — Muhimbili University of Health and Allied Sciences
Locations (2):
- Tanzania (2):
  - Kibindu, Bagamoyo, Dar esSalaam
  - Yombo Dispensary, Bagamoyo, Yombo

REFERENCES:
- [Background] Coran AG, Tyler HB. Aortic dissection. A complication of translumbar aortography. Am J Surg. 1968 May;115(5):709-11. doi: 10.1016/0002-9610(68)90107-4. No abstract available. PMID 5645671
- [Background] Smit MR, Ochomo EO, Aljayyoussi G, Kwambai TK, Abong'o BO, Chen T, Bousema T, Slater HC, Waterhouse D, Bayoh NM, Gimnig JE, Samuels AM, Desai MR, Phillips-Howard PA, Kariuki SK, Wang D, Ward SA, Ter Kuile FO. Safety and mosquitocidal efficacy of high-dose ivermectin when co-administered with dihydroartemisinin-piperaquine in Kenyan adults with uncomplicated malaria (IVERMAL): a randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2018 Jun;18(6):615-626. doi: 10.1016/S1473-3099(18)30163-4. Epub 2018 Mar 27. PMID 29602751
- [Background] Dondorp AM, Nosten F, Yi P, Das D, Phyo AP, Tarning J, Lwin KM, Ariey F, Hanpithakpong W, Lee SJ, Ringwald P, Silamut K, Imwong M, Chotivanich K, Lim P, Herdman T, An SS, Yeung S, Singhasivanon P, Day NP, Lindegardh N, Socheat D, White NJ. Artemisinin resistance in Plasmodium falciparum malaria. N Engl J Med. 2009 Jul 30;361(5):455-67. doi: 10.1056/NEJMoa0808859. PMID 19641202
- [Background] Leang R, Taylor WR, Bouth DM, Song L, Tarning J, Char MC, Kim S, Witkowski B, Duru V, Domergue A, Khim N, Ringwald P, Menard D. Evidence of Plasmodium falciparum Malaria Multidrug Resistance to Artemisinin and Piperaquine in Western Cambodia: Dihydroartemisinin-Piperaquine Open-Label Multicenter Clinical Assessment. Antimicrob Agents Chemother. 2015 Aug;59(8):4719-26. doi: 10.1128/AAC.00835-15. Epub 2015 May 26. PMID 26014949
- [Background] Mwaiswelo R, Ngasala B, Gil JP, Malmberg M, Jovel I, Xu W, Premji Z, Mmbando BP, Bjorkman A, Martensson A. Sustained High Cure Rate of Artemether-Lumefantrine against Uncomplicated Plasmodium falciparum Malaria after 8 Years of Its Wide-Scale Use in Bagamoyo District, Tanzania. Am J Trop Med Hyg. 2017 Aug;97(2):526-532. doi: 10.4269/ajtmh.16-0780. PMID 28829723
- [Background] Mwaiswelo R, Ngasala B, Jovel I, Xu W, Larsson E, Malmberg M, Gil JP, Premji Z, Mmbando BP, Martensson A. Prevalence of and Risk Factors Associated with Polymerase Chain Reaction-Determined Plasmodium falciparum Positivity on Day 3 after Initiation of Artemether-Lumefantrine Treatment for Uncomplicated Malaria in Bagamoyo District, Tanzania. Am J Trop Med Hyg. 2019 May;100(5):1179-1186. doi: 10.4269/ajtmh.18-0729. PMID 30860013